CLINICAL TRIAL: NCT00508079
Title: Incidence and Progression of Peripheral Venous Disease
Brief Title: Evaluating the Occurence of New and Progression of Existing Peripheral Venous Disease in Leg Veins
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Dr. Michael H. Criqui, Distinguished Professor, University of California, San Diego
Other Study IDs: 1389; R01HL084229-01A1 (NIH)
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Peripheral Vascular Diseases
Keywords: Venous Disease; Varicose Veins; Chronic Venous Insufficiency; PAD
MeSH Terms: conditions — Peripheral Vascular Diseases; Varicose Veins

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Peripheral venous disease occurs when a vein becomes damaged or blocked. It can occur almost anywhere in the body, but is most common in the arms and legs. This study will examine people who participated in a previous venous disease study to evaluate changes in leg veins and venous disease status over a period of 11 years.

DETAILED DESCRIPTION:
Peripheral venous disease is a general term for damage, defects, or blockage that occurs in the peripheral veins, which carry blood from the hands and feet back to the heart to receive oxygen. The most common cause of peripheral venous disease is a blood clot that blocks a vein. Varicose veins, which are swollen blood vessels near the surface of the skin, and chronic venous insufficiency, a condition in which blood in the leg veins does not drain properly, are two other common types of peripheral venous disease. From 1996 to 2000, the San Diego Population Study (SDPS) evaluated a group of individuals to gather information on the prevalence of venous disease. This current study will re-evaluate the SDPS participants to document changes that have occurred in their leg veins over the past 11 years, including any new venous disease and any progression of existing venous disease. Study researchers will also evaluate how venous disease relates to risk factors, symptoms, and quality of life issues.

This study will enroll people who participated in the SDPS study. Each participant will attend one study visit. Study staff will conduct a 1-hour interview with each participant to collect information on their medical history, disease-related symptoms, risk factors for venous disease, family health history, health habits, and quality of life. Blood collection will occur, participant's leg veins will be examined and photographed, and blood flow in the legs will be measured with an ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the SDPS study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Previous participants from the San Diego Population Study
Sampling Method: Non-Probability Sample
Enrollment: 1103 (Actual)
Dates: Start 2007-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Incident Venous Disease | Since previous visit (approximately 11 years)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H. Criqui, MD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States